CLINICAL TRIAL: NCT04475731
Title: Ponatinib for the Management of Minimal Residual Disease (MRD) and Hematologic Relapse in Adult Ph+ Acute Lymphoblastic Leukemia (Ph+ ALL) Patients
Brief Title: Ponatinib in Adult Ph+ ALL Patients With MRD Positivity or Hematological Relapse
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALL2620
Record Dates: First submitted 2020-06-25; First posted 2020-07-17 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Philadelphia-Positive ALL; Acute Lymphoblastic Leukemia, in Relapse
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — ponatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): MRD+ Ph+ ALL adult patients will receive Ponatinib x 4 weeks x 3 courses; +/-Concomitant chemotherapy (according to hematologic status).
  Patients will receive the study drug until disease relapse or progression.
  Interventions: Drug: Ponatinib

INTERVENTIONS:
Drug: Ponatinib — Ponatinib 45 mg/day x 4 weeks x 3 courses.
  +/- chemotherapy:
  * vincristine or
  * L-VAMP (leucovorin, vincristine, aracytin, methotrexate, prednisone)

SUMMARY:
This is a phase II interventional trial to evaluate if the use of ponatinib, with or without chemotherapy, can induce a molecular remission in MRD-positive patients, in patients in hematologic and extra-hematologic relapse and in the few patients who never achieved an hematologic remission after whatever prior treatment.

DETAILED DESCRIPTION:
This is a phase II interventional multicenter study for adult patients with Ph+ALL who:

* Are MRD+ (i.e. BCR-ABL1/ABL1 >0.01) (or loose their molecular response) after whichever kind of previous treatment. MRD positivity is indeed regarded as a relapse/resistance, since it represents the early recognition of cases who will eventually experience an hematologic recurrence of disease.
* Are in hematologic relapse after whichever kind of previous treatment.
* Have never achieved an hematologic remission at least after one month of treatment.

Patients will be treated with Ponatinib at a dose of 45 mg/die per os for 28 days for 3 cycles and - if in hematologic and extra-hematologic relapse/refractoriness, clinically fit and according to medical decision - with concurrent systemic chemotherapy. In case of CMR achievement, dosing will be reduced to 30 mg. In case of toxicity, Ponatinib will be reduced to 30 (or 15) mg daily.

ELIGIBILITY:
Inclusion Criteria:

1. Ph+ ALL patients with evidence of MRD disease or in hematologic and extra-hematologic relapse/refractoriness after any previous treatment, will be considered eligible to enter the study.
2. Age ≥18 years old with no upper age limit.
3. Adequate hepatic function as defined by the following criteria:

   * total serum bilirubin ≤1.5 x upper limit of normal (ULN), unless due to Gilbert's syndrome
   * alanine aminotransferase (ALT) ≤2.5 × ULN
   * aspartate aminotransferase (AST) ≤2.5 × ULN.
4. Adequate pancreatic function as defined by the following criterion:

   - serum lipase and amylase ≤1.5 × ULN.
5. For females of childbearing potential, a negative pregnancy test must be documented prior to enrollment.
6. Female and male patients who are fertile must agree to use an effective form of contraception with their sexual partners from enrollment through 4 months after the end of treatment.
7. Signed written informed consent according to ICH/EU/GCP and national local laws.

Exclusion Criteria:

1. WHO performance status ≤ 50% (Karnofsky) or ≥ 3 (ECOG).
2. Uncontrolled active HBV or HCV hepatitis, or AST/ALT ≥ 2.5 x ULN and bilirubine ≥ 1.5 x ULN not due to the disease.
3. History of acute pancreatitis within 1 year of study or history of chronic pancreatitis.
4. History of alcohol abuse.
5. Ongoing or active uncontrolled infections.
6. Uncontrolled hypertriglyceridemia (triglycerides >450 mg/dL).
7. Clinically significant, uncontrolled or active cardiovascular disease, specifically including, but not restricted to:

   * any history of myocardial infarction, stroke, or revascularization
   * unstable angina or transient ischemic attack within 6 months prior to enrollment
   * congestive heart failure within 6 months prior to enrollment, or left ventricular ejection fraction (LVEF) less than lower limit of normal per local institutional standards within 6 months prior to enrollment
   * history of clinically significant (as determined by the treating physician) atrial arrhythmia
   * any history of ventricular arrhythmia
   * any history of venous thromboembolism including deep venous thrombosis or pulmonary embolism
   * uncontrolled hypertension (diastolic blood pressure >90 mm Hg; systolic >140 mm Hg). Patients with hypertension should be under treatment on study entry to effect blood pressure control.
8. Taking medications that are known to be associated with Torsades de Pointes.
9. Taking any medications or herbal supplements that are known to be strong inhibitors of CYP3A4 within at least 14 days before the first dose of ponatinib.
10. Creatinine level >2.5mg/dl or glomerular filtration rate (GFR) <20 ml/min or proteinuria >3.5 g/day.
11. Patients who are currently receiving treatment with any of the medications listed in Appendix E if the medications cannot be either discontinued or switched to a different medication prior to starting study drug. The medications listed in Appendix E have the potential to prolong QT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2021-05-04 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
MRD negativity/reduction rate | After 3 months of treatment
  Rate of patients who achieve a MRD negativity/MRD reduction following treatment with either Ponatinib alone or in combination with systemic chemotherapy

SECONDARY OUTCOMES:
Duration of CMR | at 24 months
  Duration of the CMR status after 3 months of ponatinib treatment
Hematologic remission rate | at 24 months
  The achievement of an hematologic remission in patients treated for an hematologic and extra-hematoloigc relapse and for a refractory disease.
Best molecular response | at 24 months
  Best molecular response achieved during the follow-up
Rate of AE/SAEs | at 24 months
  Safety profile in terms of incidence of grade >3 CTC-NCI side effects and toxicities (AE/SAEs).
Mutational analysis | at 24 months
  Mutational analysis in terms of occurrence, type and number of BCR-ABL1 kinase domain mutations.
Correlation between biological and MRD parameters | at 24 months
  Correlation between the achievement and duration of CMR (or MRD reduction) with the type of fusion protein (e.g. p190 or p210) and the potential occurrence of mutations, as well as with additional genomic lesions.
Disease free survival | 24 months
  Time interval between the achievement of CHR after three months of ponatinib and hematologic relapse of the disease or death in CHR; patients still alive, in CHR.
Overall survival | 24 months
  Time interval between treatment start and death for any cause.
Cumulative incidence of relapse | 24 months
  Time interval between achievement of CHR after three months of ponatinib until the date of first hematologic relapse of the disease.
Role of hematological profile on survival outcome | at 24 months
  Identification of hematological profile on survival outcome

CONTACTS AND LOCATIONS:
Locations (22):
- Italy (22):
  - Aou Ospedali Riuniti "Umberto I - G.M. Lancisi - G. Salesi"- Ancona - Sod Clinica Ematologica, Ancona
  - Area Vasta N. 5 Ascoli Piceno - S. Benedetto Del Tronto, Presidio Ospedaliero Av5 Osp. Gen. Prov.Le "C.G.Mazzoni" - Uoc Ematologia, Ascoli Piceno
  - Ao Di Rilievo Nazionale E Di Alta Specialità "San Giuseppe Moscati" - Avellino - Uoc Ematologia Con Unità Di Trapianto, Avellino
  - Aou Consorziale Policlinico - Bari - Uo Ematologia Con Trapianto, Bari
  - Asst Papa Giovanni Xxiii - Ospedale Di Bergamo - Sc Ematologia, Bergamo
  - Aou Di Bologna - Policlinico S. Orsola-Malpighi - Uoc Ematologia, Bologna
  - Asst Degli Spedali Civili Di Brescia - Uo Ematologia, Brescia
  - Aso S. Croce E Carle - Cuneo - Sc Ematologia, Cuneo
  - Aou Careggi - Firenze - Sod Ematologia, Florence
  - Aou Policlinico "G. Martino" - Messina - Uoc Ematologia, Messina
  - Aulss 3 Serenissima, Ospedale Dell'Angelo - Mestre - Uo Ematologia, Mestre
  - Asst Grande Ospedale Metropolitano Niguarda - Milano - Sc Ematologia, Milan
  - Irccs Ospedale S. Raffaele - Milano - Uo Oncoematologia, Milan
  - Aou Federico Ii - Napoli - Uoc Ematologia, Napoli
  - Ao Di Perugia, Ospedale S. Maria Della Misericordia - Ematologia E Trapianto Midollo Osseo, Perugia
  - Ao Ospedali Riuniti Marche Nord - Ospedale San Salvatore - Pesaro - Uoc Ematologia E Centro Trapianti, Pesaro
  - Università Degli Studi Di Roma "Sapienza" - Dipartimento Di Medicina Traslazionale E Di Precisione - U.O.C. Ematologia, Roma
  - Aou "San Giovanni Di Dio E Ruggi D'Aragona" - Salerno - Uoc Ematologia E Trapianti Di Cellule Staminali Emopoietiche, Salerno
  - Ente Ecclesiastico Casa Sollievo Della Sofferenza - San Giovanni Rotondo - Ematologia, San Giovanni Rotondo
  - Aou Senese - Uoc Ematologia E Trapianti, Siena
  - Aou Città Della Salute E Della Scienza, Ospedale S. Giovanni Battista Molinette - Torino - Sc Ematologia 2, Torino
  - Aou Integrata Di Verona, Policlinico G.B. Rossi - Uoc Ematologia, Verona